CLINICAL TRIAL: NCT04469309
Title: Comparison of Half-Somersault Exercise With Brandt-Daroff Exercise in Patients With Posterior Canal Benign Paroxysmal Positional Vertigo: A Randomized Clinical Trial
Brief Title: Comparison of Half-Somersault Exercise With Brandt-Daroff Exercise in BPPV.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00744 M Jaffar
Record Dates: First submitted 2020-04-14; First posted 2020-07-14 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Vertigo, Paroxysmal
Keywords: Half-Somersault Exercise; Brandt-Daroff exercise; Posterior Canal; Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Vertigo; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Group I will receive Brandoff Exercises
  Interventions: Other: Group I Brandt-Daroff Exercises
- Group II (Active Comparator): Group II will receive Somersault exercises
  Interventions: Other: Group II Half-Somersault Maneuver

INTERVENTIONS:
Other: Group I Brandt-Daroff Exercises — In group I Brandoff Exercises will be performed using standard method, in which the patient is in the sitting position on examination table, the patient moves into the lying position on the affected side on the shoulder, with the head angled upward with about 45. The patient stays in this for 30 s and then goes back to the sitting position, looks forward and remains in this position for 30 s as well. The patient repeats the same procedure for the other side, too.
  The patient performs this maneuver 2 times, twice a day. For total 9 days for 3 weeks. Pre, mid and post assessment.
  Arms: Group I
Other: Group II Half-Somersault Maneuver — In group II Half-Somersault Maneuver will be done, the patient performs this maneuver 2 times, twice a day. For total 9 days for 3 weeks.
  Arms: Group II

SUMMARY:
This study is important as there are numbers of BPPV patients presenting to outpatient departments which needs more efficient techniques for management of BPPV. Talking about literature, there are numbers of studies done on different maneuvers but there is yet no study available which compares these maneuvers. So the purpose of this study is to compare these techniques to find which one is more effective in treating PC-BPPV.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is one of the most common causes in patients with vestibular disorders .BPPV has often been described as "self-limiting" because symptoms often subside or disappear within six months of onset . BPPV may be characterized by sudden changes in the position of the head, such as lying down on one or both sides, looking right or left side . Vertigo is defined as illusion of movement which could be spinning, rocking, tilting or dropping . Benign paroxysmal positional vertigo (BPPV) is the most frequent vestibular disorder and the leading cause of vertigo in adults.BPPV may be divided into 3 types based on canal involvement i.e Posterior, Horizontal, and Anterior Semicircular Canal BPPV. BPPV clinical findings agree with the hypothesis that semicircular canals with greater incidence is posterior canal, have floating particles or debris, which are heavier than the circulating endolymph . The vestibular system is located in the inner ear and consists of the utricle, saccule and three semicircular canals (i.e. posterior, anterior and horizontal). These canals react to rotational movements of the head . Of the types of BPPV, posterior semicircular canal BPPV (PC-BPPV) is the most common form, accounting for 85 to 90% of cases Lateral Canal BPPV is about 20%, and Anterior Canal BPPV is very rare as it is self-treated due to gravity . BPPV accounts for 8% of the subjects with moderate or severe dizziness/vertigo. It may be present in child hood but increases with age. The lifetime prevalence is estimated to be 2%. It´s reported that the oneyear prevalence is 0.5% in 18-39 years old and 3.4% in people over 60-years of age . Benign paroxysmal positional vertigo (BPPV) is the paroxysmal transient vertigo caused by specific changes in head position, accounting for 60% of peripheral vertigo, with an incidence rate of approximately 64/10000 . The average recurrence rate is around 50%. BPPV is more common in women than men; and the ratio of women to man population is 2:1.BPPV can be caused either by canalithiasis or by cupulolithiasis. Movement of the head causes these otoliths to inappropriately trigger the receptors in the semicircular canals and send false signals to the brain, causing vertigo and nystagmus . Factors that can be helpful in guiding the clinician in the evaluation of the patient with dizziness include the characteristics of the dizziness; associated symptoms (ie, hearing loss or tinnitus) duration of symptoms; and what, if anything, triggered the symptoms (precipitating factors) . Posterior canal BPPV is treated using canalith repositioning procedures, the most common of which is the Epley maneuver(EM) , half somersault exercises , Brandt Daroff exercise , Semont maneuver, vestibular habituation exercises, balance and eye exercises . Dix-Hallpike test is used to diagnose BPPV patients . Paramasivan Mani et al suggested in their study that half somersault exercise with Brandt Daroff exercise for 3 weeks showed significantly greater improvement in reducing self-perceived handicap among Patients with Posterior Canal Benign Paroxysmal Positional Vertigo . Ashok Kumar Gupta et.al concluded that Epley maneuver has produced maximum improvement than Semont maneuver and least improvement was produced by Brandt-Daroff Exercises . Herman Guild Manayil John et al observed in their study that Epley's manoeuvre to be a simple, useful and cost-effective treatment for BPPV . Nevzat Demirbilek, conducted a study of Combined Epley and Semont Maneuver in Benign Paroxysmal Positional Vertigo and concluded that, the combined maneuvers in our study were found to have an increased success rate . Devangi S. Desai et al concluded that, both Epley's maneuver and Brandt-daroff treatment approaches are effective in reducing symptoms and improving independence level but combined approaches can give better results so modified epley'smaneuver should be applied 3 times in one session along with brandt- daroff exercise as home exercise .

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Patients with PC-BPPV
* Age group 25-50 years.
* DHI Scale: 36-42 (moderate handicap)
* Both gender
* Duration of complaints: from the past 6 months

Exclusion Criteria:

* Migraine related dizziness and Anxiety disorder
* Other vestibular conditions are: Acoustic neuroma, Labyrinthitis, Vestibular hypo function, Meniere's disease.
* Any cervical pathology,
* CNS Pathology causing dizziness and vertigo
* Other pathologies which may affect balance.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Vestibular activities and participation measure | Change from Baseline dizziness and balance to 2 Weeks
  The Vestibular Activities and Participation Measure (VAP) is a 34-item self-report questionnaire that asks the individual to evaluate the effect of dizziness and/or balance problems on their ability to perform activity and participation tasks.The response range from none (0 points) ,moderate (2 points), severe (3 points) unable to do (4 points) to not applicable. The total score is obtained after calculating the average of the item scale values and excluding the not applicable item scale scores
Dix-Hall pike test | Change from Baseline dizziness to 2 Week
  Dix-Hall pike is the standard procedure for diagnosis of PC-BPPV. The Dix-Hallpike Test (DHT) is considered the gold standard assessment for the diagnosis of the vestibular disorder Benign Paroxysmal Positional Vertigo (BPPV). The Dix-Hallpike test involves rapidly moving the patient from a sitting position to "head hanging," where the patient's head is at least 10 degrees below horizontal.

SECONDARY OUTCOMES:
Fall efficacy scale (FES) | Change from Baseline dizziness to 2 Week
  Fall efficacy scale (FES) scale is a measure used to quantify an individual's concern of falling during different tasks. The FES is a reliable and valid tool for measuring an individual's concern of falling in a sample of people with vestibular disorders. It consists of 10 activities which are asked from patients.On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, A total score of greater than 70 indicates that the person has a fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- HMC Hospital Peshawar, Peshawar, Khyber Pakhtunkha, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta AK, Sharma KG, Sharma P. Effect of Epley, Semont Maneuvers and Brandt-Daroff Exercise on Quality of Life in Patients with Posterior Semicircular Canal Benign Paroxysmal Positional Vertigo (PSCBPPV). Indian J Otolaryngol Head Neck Surg. 2019 Mar;71(1):99-103. doi: 10.1007/s12070-018-1322-7. Epub 2018 Mar 30. PMID 30906723
- [Background] Maranhao ET, Whitney SL, Maranhao-Filho P. Tumarkin-like phenomenon as a sign of therapeutic success in benign paroxysmal positional vertigo. Arq Neuropsiquiatr. 2018 Aug;76(8):534-538. doi: 10.1590/0004-282X20180073. PMID 30231127
- [Background] Beeumen N Van. Faculteit Geneeskunde en Levenswetenschappen master in de revalidatiewetenschappen en de kinesitherapie Faculteit Geneeskunde en Levenswetenschappen master in de revalidatiewetenschappen en de kinesitherapie. 2018
- [Background] Zhang YX, Wu CL, Zhong FF, Ding CN. Evaluation of efficacies and recurrence rates of three self-treatment maneuvers for posterior semicircular canal benign paroxysmal positional vertigo. Int J Clin Exp Med. 2016;9(6):11780-7
- [Background] Kinne BL. Benign paroxysmal positional vertigo. Eye Mov Disord (Nystagmus Strabismus) Diagnosis, Manag Impact Qual Life. 2014;9(1):1-30.
- [Background] Desai DS, Chauhan AS, Trivedi MN. Role of Modified Epley'S Maneuver and Brandt-Daroff Exercises in Treatment of Posterior Canal Bppv: a Comparative Study. Int J Physiother Res. 2015;3(3):1059-64.
- [Background] Manayil John HG, John A. Efficacy of Epley'S Manoeuvre in Posterior Canal Benign Paroxysmal Positional Vertigo. J Evid Based Med Healthc. 2016;3(102):5624-7.
- [Derived] Jaffar M, Ghous M, Ayaz M, Khan AA, Akbar A, Haleem F. Effects of Half-Somersault and Brandt-Daroff exercise on dizziness, fear of fall and quality of life in patients with posterior canal benign paroxysmal positional vertigo: A randomised control trial. J Pak Med Assoc. 2023 Jan;73(1):139-142. doi: 10.47391/JPMA.3333. PMID 36842024